CLINICAL TRIAL: NCT04029376
Title: Non-Interventional Study of Children Aged From 3 to 14 Years Suffering From Functional Gastrointestinal Complaints Classified According to the Rome Criteria
Brief Title: Study to Learn More About the Stomach and Intestine Complaints of Children Aged From 3 to 14 Years
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 20983
Record Dates: First submitted 2019-07-22; First posted 2019-07-23 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Functional Gastrointestinal Disorders
MeSH Terms: conditions — Gastrointestinal Diseases | interventions — iberogast

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Iberogast® — The medication was applied 3 times 20 drops per day before or at meals with some liquid, ideally to one week insofar.

SUMMARY:
In this observational study, researchers want to gain more information on children suffering from abnormal stomach and intestine function (based on the Rome criteria) and treated Iberogast. The Rome criteria have been developed by experts to support doctors to diagnose stomach and intestine disorders. This study will focus on children aged from 3 to 14 years in age treated by their doctor with the herbal drug Iberogast for their stomach and intestine complaints for one week. Researcher want to learn more about the efficacy of Iberogast by observing the changes of symptoms related to the stomach and intestine disorders. In addition information on the safety of the drug and how well the drug is tolerated by the patients will be collected.

ELIGIBILITY:
The selection of the children to be documented was the sole responsibility of the physician whereby the information of the Rome III criteria on functional gastrointestinal diseases in children as well as the prescribing information on Iberogast could be consulted as guideline. Only the therapeutic necessity was determining for the use of all medicines. The treating physicians received standardised information regarding the ailment picture (Rome III criteria) before the beginning of the study and during the investigator meetings.

Ages: 3 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Male and female children aged between 3 and up to 14 years with Functional Gastrointestinal Complaints
Sampling Method: Probability Sample
Enrollment: 1032 (Actual)
Dates: Start 2007-04-01 (Actual); Primary Completion 2008-10-01 (Actual); Study Completion 2008-10-01 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal Symptoms Profile (GIS) Score | Up to 1 week
  The score was developed by Steigerwald Arzneimittelwerk GmbH in co-operation with a gastroenterological expert group and validated (Holtmann et al. 2004, Adam et al., 2005). It consists of 10 individual symptoms that were regarded as being typical for dyspepsia. They were evaluated based on a 5-stage Likert scale. The score was adapted to the special situation of children and adolescents with functional gastrointestinal disorders as part of the study concept. The change in the summary score during therapy serves as evaluation criterion for the efficacy of the therapeutic measure. The symptoms profile essentially involves all the symptoms of functional dyspepsia mentioned by the German Society for Gastrointestinal and Metabolic Diseases (DGVS) or international Rome criteria. Its usability was confirmed by the validation procedure.
Global Assessment of the Efficacy by the Physicians | Up to 1 week
  Treatment success assessed by physicians
Global Assessment of the Efficacy by the Children or Their Parents | Up to 1 week
  Treatment success judged by children or their parents
Lost Attendance days | Up to 1 week
  The number of lost attendance days kindergarten/school

SECONDARY OUTCOMES:
Global Assessment of the Tolerability by the Physician | Up to 1 week
  The tolerability of Iberogast assessed by physician
The number of subjects with adverse events | Up to 1 week
  The number of subjects who had any adverse event during the study

CONTACTS AND LOCATIONS:
Locations (1):
- Many locations, Multiple Locations, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com/